CLINICAL TRIAL: NCT00524953
Title: Phase I - Clinical Trial to Assess Safety of Ultraviolet (UV) Phototherapy for the Prevention of Graft Versus Host Disease After Allogeneic Stem Cell Transplantation
Brief Title: Phase I Clinical Trial to Assess Safety of UV Phototherapy for the Prevention of GVHD Post Allogeneic SCT
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UV-GVHD - HMO-CTIL
Record Dates: First submitted 2007-09-04; First posted 2007-09-05 (Estimated); Last update posted 2015-06-11 (Estimated); Status verified 2007-08

CONDITIONS: Allogeneic Transplantation (Non T-cell Depleted)
Keywords: allogeneic bone marrow transplantation; non-T-cell depleted; UV-c; GVHD

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- I (Experimental): 10 patients after allogeneic BMT (non T-depleted).
  Interventions: Device: EUMATRON - EN 600 NT

INTERVENTIONS:
Device: EUMATRON - EN 600 NT — frequency - once a week, starting 4 days after transplantation for four weeks (total of 4 treatments) each treatment will last ~20 minutes. In addition - standard GVHD preventive protocol will be given to patients (including cyclosporine and steroids - if necessary)
  Other Names: EN 600 NT

SUMMARY:
The primary goal of thos study is to assess safety of Ultraviolet (UV) Phototherapy for the Prevention of Graft versus Host Disease after allogeneic stem cell transplantation (Phase I - Clinical trial). Following allogeneic BMT, patients will be placed on standard GVHD preventive therapy (cyclosporine).

Secondary goals -

* monitoring immune system recovery
* the influence of stem cells origin on therapy and/orGVHD prevention
* the influence of UV-c treatment on survival

clinical data and samples will be collected, during UV-c therapy, 100 days after discharge & 6 months after discharge - to examine the long-term effect of UV-c treatment on the patient's GVHD status.

DETAILED DESCRIPTION:
Treatment will be given with a portable, easy to operate device named "EUMATRON". this device contains a UV- lamp. 250 cc of blood from a peripheric vein is going through the device into a bottle with Low dose Heparin and returning to patient's body. procedure takes ~20 minutes.

ELIGIBILITY:
Inclusion Criteria:

* patients post non T cell depleted allogeneic stem cell transplantation

Exclusion Criteria:

* morbidity unrelated to GVHD
* patients in an hemodynamic unstable condition
* acute uncontrolled bleeding
* patients undergoing dialysis

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-09; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
safety and tolerability of UV-c phototherapy for the Prevention of Graft versus Host Disease after allogeneic stem cell transplantation | 6 months

SECONDARY OUTCOMES:
monitoring immune system recovery, influence on survival rates, influence of stem cells origin on treatment & prevention of GVHD | 100 days, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Reuven Or, MD, Principal Investigator — Bone Marrow transplantation, cancer immunotherapy & immunobiology research center, Hadassah University Hospital, Ein - Kerem, Jerusalem, Israel
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel